CLINICAL TRIAL: NCT06447246
Title: Respiratory Effects of Obesity in Children: Longitudinal Consequences After 6 Years of Aging
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Tony Babb, PROFESSOR, Cardiopulmonary Laboratory Director, Effie and Wofford Cain Chair in Cardiopulmonary Research, Institute of Exercise and Environmental Medicine, Division of Pulmonary and Critical Care Medicine, University of Texas Southwestern Medical Center
Other Study IDs: STU-2024-0444; 5R01HL136643-05 (NIH)
Record Dates: First submitted 2024-05-29; First posted 2024-06-07 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Children With Obesity: No intervention or treatment will be administered. This group will not return after initial visits.
- Children Without Obesity: No intervention or treatment will be administered. This group will not return after initial visits.

SUMMARY:
The purpose of the study is to re-examine body composition, respiratory function, exercise tolerance, and dyspnea on exertion (DOE) in children with obesity (CWO) and children without obesity (CWOO) who were originally studied as 8-12-year-olds between 2016-2023 (i.e., originally Tanner score ≤ 3; 90 participants; 26 CWOO & 64 CWO).

DETAILED DESCRIPTION:
The prevalence of childhood obesity increases with age (20.7% aged 6-11 & 22.2% aged 12-19; NHANES 2017-2020). CWO, compared with CWOO, are more likely to have chronic health conditions.

Results from the investigator's prior grant (HL136643) show that over one year, CWO can add four times as much fat weight as CWOO. However, it is unknown if this rate of increase in fat weight continues into adolescence and early adulthood, and whether respiratory function, exercise tolerance, or DOE are progressively worsened by increasing obesity. Furthermore, there could be a sex difference in the effects of obesity, given the different growth characteristics for boys and girls.

The investigator's long-term objective is to investigate the effects of 6 years of aging on body composition, respiratory function, exercise tolerance, and DOE in CWO and CWOO.

Specific Aims: The investigators will test the following hypotheses in CWO and CWOO after 6 years of aging:

Aim 1) CWO originally studied at 8-12 years old will demonstrate a greater increase in fat weight and lower respiratory function (i.e., altered pulmonary function & breathing mechanics at rest) than in CWOO originally studied at 8-12 years old;

Aim 2) CWO originally studied at 8-12 years old will demonstrate lower exercise tolerance measured during graded cycle ergometry (as evidenced by peak V • O2 in ml/min/kg, i.e., physical fitness) than in CWOO originally studied at 8-12 years old, but not lower cardiorespiratory fitness (as evidenced by peak V • O2 in % of predicted based on ideal body wt., i.e. cardiorespiratory fitness);

Aim 3) CWO originally studied at 8-12 years old will demonstrate greater DOE as evidenced by increased ratings of perceived breathlessness during constant load exercise cycling than in CWOO originally studied at 8-12 years old; and

ELIGIBILITY:
Inclusion Criteria:

The participants originally studied as 8-12-year-olds between 2016-2023 as part of the investigator's R01 HL136643.

Exclusion Criteria:

1. Children not able to follow directions, adequately perform procedures (e.g., pulmonary function tests), or keep appointments (e.g., no shows for testing).
2. If a child developed an abnormal ECG, showed other signs of clinical exercise intolerance, or signs of cardiovascular/lung disease during the exercise test, testing was terminated, and the child was referred to their personal physician for further evaluation.
3. Women who are pregnant or could possibly be pregnant (i.e. not using approved birth control measures and sexually active) will be excluded because of changes in body size during pregnancy and because unforeseeable risks to the fetus.
4. Presence of significant disease defined as a disease which in the opinion of the investigator may put the subject at risk because of participation in the study or a disease that may influence the results of the study or the subject's ability to participate in the study.
5. Patients who are non-English speaking will be excluded from the study because the tests performed are very effort dependent, detailed and require technical communication between the staff and the patient. The investigators feel that a translator would not be able to translate the technical terms fast enough to instruct the patient in the testing.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The participants originally studied as 8-12-year-olds between 2016-2023 as part of the investigator's R01 HL136643.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-08-23 (Actual); Primary Completion 2029-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Pulmonary Function: Lung Volumes | Change from Baseline in differences between nonobese and obese children. Outcome measures will be assessed within 48-72 hours after completion of each study.
  Pulmonary function is comprised of several physiological variables but this study will primarily measure Lung Volume: FRC (liters) and TLC (liters)
Exercise Tolerance - Peak VO2 | Change from Baseline in differences between nonobese and obese children. Outcome measures will be assessed within 48-72 hours after completion of each study.
  Exercise Tolerances is represented by several physiological variables but the primary variable is Maximal oxygen uptake (L/min and percent predicted)
Dyspnea on Exertion | Change from Baseline in differences between nonobese and obese children. Outcome measures will be assessed within 48-72 hours after completion of each study.
  Dyspnea on Exertion is represented using the Borg Scale which provides Ratings of Perceived Breathlessness (RPB) during constant load exercise cycling. The Borg Scale measures from 0-10, where 0 = no breathlessness and 10 = maximal breathlessness.

OTHER OUTCOMES:
Pulmonary Function: Spirometry | Change from Baseline in differences between nonobese and obese children. Outcome measures will be assessed within 48-72 hours after completion of each study.
  Spirometry includes: Forced vital capacity (% predicted), Forced Expiratory Volume in 1 second (FEV1) (% predicted), FEV1/FVC (% predicted), and peak flow (% predicted.)
Pulmonary Function: Diffusing Capacity | Change from Baseline in differences between nonobese and obese children. Outcome measures will be assessed within 48-72 hours after completion of each study.
  Diffusing Capacity: Diffusing capacity of lung for carbon monoxide(DLco) (ml/mmHg/min)
Exercise Tolerance: Work Rate | Change from Baseline in differences between nonobese and obese children. Outcome measures will be assessed within 48-72 hours after completion of each study.
  Associated variables such as work rate (W)
Exercise Tolerance: Minute Ventilation | Change from Baseline in differences between nonobese and obese children. Outcome measures will be assessed within 48-72 hours after completion of each study..
  Associated variables such as pulmonary ventilation (L/min)
Exercise Tolerance: Operational Lung Volumes | Change from Baseline in differences between nonobese and obese children. Outcome measures will be assessed within 48-72 hours after completion of each study.
  Associated variables such as operational lung volumes (EELV and EILV as a % of TLC)

CONTACTS AND LOCATIONS:
Overall Officials: Tony G Babb, Ph.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Institute for Exercise and Environmental Medicine, UT Southwestern and Texas Health Presbyterian Hospital Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No